CLINICAL TRIAL: NCT03820726
Title: An Open-label Extension Trial of the Long Term Safety of Nintedanib in Patients With Progressive Fibrosing Interstitial Lung Disease (PF-ILD)
Brief Title: A Follow-up Study Investigating Long Term Treatment With Nintedanib in Patients With Progressive Fibrosing Interstitial Lung Disease (PF-ILD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199-0248; 2018-000525-32 (EudraCT Number)
Record Dates: First submitted 2019-01-28; First posted 2019-01-29 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nintedanib (Experimental): Patients taking 150 milligram (mg) bid blinded trial medication (active drug or placebo) at the end of INBUILD® started treatment with nintedanib 150 mg bid in this extension trial. Patients taking 100 mg bid blinded trial medication (active drug or placebo) at the end of INBUILD® started treatment with nintedanib in this extension trial either at 100 mg bid or at an increased dose of 150 mg bid at the discretion of the investigator orally as soft gelatine capsule, twice daily (bid), together with a glass of water (~250 mL), in a dose interval of 12 hours. With an optional dose reduction to 100 mg bid temporarily or permanently to manage adverse events (AEs). The treatment had a duration of 96 weeks or until nintedanib was made available to the patients outside of the clinical trial. Treatment was stopped if any reason for withdrawal was met.
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Bid

SUMMARY:
The main objective is to assess long term tolerability and safety of treatment with oral nintedanib in patients with Progressive Fibrosing Interstitial Lung Disease (PF-ILD) who have complete (and did not prematurely discontinue trial medication in) the phase III parent trial, INBUILD® (trial 1199.247).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who completed the INBUILD® trial as planned and who did not prematurely discontinue blinded treatment.
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
* Women of childbearing potential (WOCBP)1 must continue to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly, as well as one barrier method, for 28 days prior to and 3 months after nintedanib administration. A list of contraception methods meeting these criteria is provided in the patient information

Exclusion Criteria:

* Any disease that may put the patient at risk when participating in this trial. Reconsider carefully all exclusion criteria of the INBUILD® trial. However, patients may qualify for participation even though exclusion criteria may have been met during the course of participation in INBUILD®, if the investigator's benefit-risk assessment remains favourable.
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Patient not compliant in parent trial (INBUILD®), with trial medication or trial visits, according to investigator's judgement.
* Previous enrolment in this trial. Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (121):
- United States (33):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis, Sacramento, California
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Pulmonary and Sleep of Tampa Bay, Brandon, Florida
  - University of Florida College of Medicine, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Pulmonary and Critical Care Associates of Baltimore, Towson, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Creighton University, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
  - NewYork-Presbyterian/Weill Cornell Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Oregon Clinic, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Medical Arts and Research Center (MARC), San Antonio, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Inova Fairfax Medical Campus, Falls Church, Virginia
- Argentina (5):
  - Centro Dr. Lazaro Langer S.R.L, Alberdi Sur
  - Centro de Investigaciones Metabólicas (CINME), C.a.b.a
  - CEMER-Centro Medico De Enfermedades Respiratorias, Florida
  - INSARES, Mendoza
  - Instituto Médico de la Fundación Estudios Clínicos, Rosario
- Belgium (4):
  - ULB Hopital Erasme, Brussels
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
  - Yvoir - UNIV UCL de Mont-Godinne, Yvoir
- Canada (4):
  - Winnipeg Clinic, Winnipeg, Manitoba
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - CHUS Fleurimont, Sherbrooke, Quebec
- Chile (3):
  - Hospital Clínico Reg. de Concepción "Dr. G. Grant Benavente", Concepción
  - Instituto Nacional del Tórax, Providencia, Santiago de Chile
  - Centro de Investigación del Maule, Talca
- China (3):
  - Peking Union Medical College Hospital, Beijing
  - Nanjing Drum Tower Hospital, Nanjing
  - The First Hospital of China Medical University, Shenyang
- France (12):
  - HOP Avicenne, Bobigny
  - HOP Louis Pradel, Bron
  - HOP Côte de Nacre, Caen
  - CHRU Lille, Lille
  - HOP Nord, Marseille
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP Pasteur, Nice
  - HOP Bichat, Paris
  - HOP Maison Blanche, Reims
  - HOP Pontchaillou, Rennes
  - HOP Civil, Strasbourg
  - HOP Bretonneau, Tours
- Germany (7):
  - Universitätsklinikum Bonn AöR, Bonn
  - Fachkrankenhaus Coswig GmbH, Coswig
  - Klinik Donaustauf, Donaustauf
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Petrus-Krankenhaus, Wuppertal
- Italy (6):
  - A.O.U. Policlinico Vittorio Emanuele, Catania
  - Ospedale "G.B. Morgagni - L. Pierantoni" ausl forli, Forlì
  - Azienda Ospedaliera Policlinico di Modena, Modena
  - A.O. San Gerardo di Monza, Monza
  - Poli Univ A. Gemelli, Roma
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
- Japan (17):
  - Tosei General Hospital, Aichi, Seto
  - Kurume University Hospital, Fukuoka, Kurume
  - Sapporo Medical University Hospital, Hokkaido, Sapporo
  - National Hospital Organization Himeji Medical Center, Hyogo, Himeji
  - Kobe City Medical Center General Hospital, Hyogo, Kobe
  - Ibarakihigashi National Hospial, Ibaraki, Naka-gun
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Tohoku University Hospital, Miyagi, Sendai
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Osaka, Sakai
  - Osaka Medical College Hospital, Osaka, Takatsuki
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
  - Tokushima University Hospital, Tokushima, Tokushima
  - Tokyo Medical and Dental University Hospital, Tokyo, Bunkyo-ku
  - Toranomon Hospital, Tokyo, Minato-ku
  - JR Tokyo General Hospital, Tokyo, Shibuya-ku
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo, Shinjuku-ku
- Poland (5):
  - University Clinical Center, Gdansk, Gdansk
  - Leszek Giec Upper-Silesian Med.Cent.Silesian Med.Univ., Katowice
  - Norbert Barlicki University Clinical Hospital No.1, Lodz, Lodz
  - Nat.Instit.of Tuberculosis&LungDiseases,Outpat.Clin,warszawa, Warsaw
  - Clinical Hospital No. 1, n.a. Prof. Szyszko from Silesian MA, Zabrze
- Russia (5):
  - Res.Inst.-Compl.Iss.Cardi.Dis., Kemerovo
  - Central Scientific Research Insitute of Tuberculosis, Moscow
  - Moscow 1st State Med.Univ.n.a.I.M.Sechenov, Moscow
  - 1stPavlov St.Med.Univ.St.-Petersburg Res.Inst., Saint Petersburg
  - Emergency Clinical Hospital n. a. N. V. Solovyev, Yaroslavl, Yaroslavl
- South Korea (3):
  - The Catholic University of Korea, Bucheon St.Mary's Hospital, Bucheon-si
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
- Spain (8):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital de Galdakao, Galdakao
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - Hospital La Princesa, Madrid
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Espases, Palma de Mallorca
  - Hospital de Canarias, San Cristóbal de La Laguna
  - Hospital Virgen del Rocío, Seville
- United Kingdom (6):
  - Royal Infirmary of Edinburgh, Edinburgh
  - St James's University Hospital, Leeds
  - Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester
  - University Hospital Llandough, Penarth
  - Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame frame' are fulfilled , researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Wuyts WA, Bonella F, Chaudhuri N, Varone F, Antin-Ozerkis D, Song JW, Miede C, Dumistracel M, Coeck C, Cottin V. Continued Treatment with Nintedanib in Patients with Progressive Pulmonary Fibrosis: Data from INBUILD-ON. Lung. 2025 Jan 9;203(1):25. doi: 10.1007/s00408-024-00778-z. PMID 39789408
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A phase III, open label, extension trial. The study aimed to evaluate the long-term tolerability and safety of oral nintedanib treatment in patients with Progressive Fibrosing Interstitial Lung Disease (PF-ILD) who have completed (and did not prematurely discontinue trial medication in) the phase III parent trial, 1199.247 (INBUILD®) NCT02999178.
Pre-assignment Details: Only patients with PF-ILD who completed the parent trial (INBUILD®) on treatment (i.e., did not discontinue treatment early) were eligible and were included in this trial if they fulfilled all the inclusion criteria and did not present any of the exclusion criteria.
Period: Overall Study
Arm/Group | Nintedanib
Started | 435
Treated | 434
Completed (Completed planned treatment period) | 224
Not Completed | 211
Not completed — Other than listed | 23
Not completed — Withdrawal by Subject | 37
Not completed — Lost to Follow-up | 3
Not completed — Protocol deviation | 1
Not completed — Adverse Event | 146
Not completed — Not treated | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This set included all patients who were dispensed trial medication (nintedanib) and were documented to have taken at least 1 dose of open-label trial medication (nintedanib).
Arm/Group | Nintedanib
Number analyzed (Participants) | 434
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211
  Male | 223
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 65
  Not Hispanic or Latino | 328
  Unknown or Not Reported | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 108
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 279
  More than one race | 1
  Unknown or Not Reported | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events
Description: Number of participants with adverse events over the course of the extension trial, AEs defined as any untoward medical occurrence in a patient administered with the investigational product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: From first nintedanib intake until last nintedanib intake + 28 days of Residual effect period (REP), up to 1195 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib
Number analyzed (Participants) | 434
Participants | 417

ADVERSE EVENTS:
Time Frame: From first nintedanib intake until last nintedanib intake + 28 days of Residual effect period (REP), up to 1195 days.
Description: Treated Set (TS): This set included all patients who were dispensed trial medication (nintedanib) and were documented to have taken at least 1 dose of open-label trial medication (nintedanib).
Arm/Group | Nintedanib
All-Cause Mortality (participants affected / at risk) | 83/434
Serious Adverse Events (participants affected / at risk) | 234/434
Other Adverse Events (participants affected / at risk) | 371/434
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=434)
Leukocytosis (Blood and lymphatic system disorders) | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 7
Atrial flutter (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 4
Cardiac failure (Cardiac disorders) | 7
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 5
Cor pulmonale chronic (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 3
Pericarditis (Cardiac disorders) | 1
Prinzmetal angina (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 1
Sinus arrest (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Age-related macular degeneration (Eye disorders) | 1
Cataract (Eye disorders) | 2
Diplopia (Eye disorders) | 1
Glaucoma (Eye disorders) | 2
Normal tension glaucoma (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Faecaloma (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Melaena (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 2
Pneumatosis intestinalis (Gastrointestinal disorders) | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3
Small intestinal obstruction (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 3
Chest pain (General disorders) | 4
Death (General disorders) | 4
Disease progression (General disorders) | 5
General physical health deterioration (General disorders) | 1
Impaired healing (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 2
Pyrexia (General disorders) | 2
Sudden death (General disorders) | 2
Biliary colic (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 2
Drug-induced liver injury (Hepatobiliary disorders) | 3
Gallbladder rupture (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic cytolysis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Liver injury (Hepatobiliary disorders) | 2
Abscess limb (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Appendicitis perforated (Infections and infestations) | 1
Atypical mycobacterial pneumonia (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 4
COVID-19 (Infections and infestations) | 12
COVID-19 pneumonia (Infections and infestations) | 7
Chronic tonsillitis (Infections and infestations) | 1
Coronavirus infection (Infections and infestations) | 1
Cytomegalovirus viraemia (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Enterococcal sepsis (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 3
Peritonitis (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 36
Pneumonia aspiration (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 4
Pneumonia pneumococcal (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 5
Sepsis (Infections and infestations) | 4
Septic shock (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 4
Accidental overdose (Injury, poisoning and procedural complications) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 2
Poisoning (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Liver function test increased (Investigations) | 1
Oxygen consumption increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 3
Abnormal loss of weight (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 2
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 2
Cerebral ischaemia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 5
Ischaemic stroke (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Mental impairment (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 3
Vascular parkinsonism (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 1
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Calculus urinary (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
IgA nephropathy (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Pulmonary renal syndrome (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 15
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 35
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 9
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 20
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 14
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 17
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1
Air embolism (Vascular disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Extremity necrosis (Vascular disorders) | 1
Neurogenic shock (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Vein disorder (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=434)
Abdominal pain (Gastrointestinal disorders) | 29
Abdominal pain upper (Gastrointestinal disorders) | 22
Constipation (Gastrointestinal disorders) | 23
Diarrhoea (Gastrointestinal disorders) | 256
Nausea (Gastrointestinal disorders) | 75
Vomiting (Gastrointestinal disorders) | 54
Bronchitis (Infections and infestations) | 48
COVID-19 (Infections and infestations) | 22
Nasopharyngitis (Infections and infestations) | 38
Respiratory tract infection (Infections and infestations) | 25
Urinary tract infection (Infections and infestations) | 28
Alanine aminotransferase increased (Investigations) | 43
Aspartate aminotransferase increased (Investigations) | 37
Gamma-glutamyltransferase increased (Investigations) | 31
Weight decreased (Investigations) | 69
Decreased appetite (Metabolism and nutrition disorders) | 45
Arthralgia (Musculoskeletal and connective tissue disorders) | 24
Back pain (Musculoskeletal and connective tissue disorders) | 30
Headache (Nervous system disorders) | 31
Cough (Respiratory, thoracic and mediastinal disorders) | 73
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 61
Productive cough (Respiratory, thoracic and mediastinal disorders) | 25
Hypertension (Vascular disorders) | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT03820726/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT03820726/SAP_001.pdf